CLINICAL TRIAL: NCT05647096
Title: Safety, Tolerability and Performance of the NucleoCapture Extracorporeal Therapeutic Apheresis Device in the Reduction of Circulating CfDNA/NETs in Subjects with Sepsis
Brief Title: Safety, Tolerability and Performance of the NucleoCapture Device in the Reduction of Circulating CfDNA/NETs in Subjects with Sepsis
Acronym: NUC-CAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Santersus AG (Industry)
Collaborators: ISS AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAN/01/2022
Record Dates: First submitted 2022-12-03; First posted 2022-12-12 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Sepsis; Respiratory Failure
Keywords: Sepsis; Respiratory failure
MeSH Terms: conditions — Sepsis; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the interventional treatment arm (SOC plus NucleoCapture) or the SOC treatment arm in a 2:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NucleoCapture Treatment (Experimental): Participants in the NucleoCapture treatment arm will receive Standard of Care plus three treatment sessions with the NucleoCapture treatment device. The device consists of 100ml NucleoCapture selective adsorber.
  Interventions: Device: NucleoCapture device
- Standard of Care (No Intervention): Participants in the Standard of Care arm will receive standard medical care alone.

INTERVENTIONS:
Device: NucleoCapture device — 100ml NucleoCapture selective DNA adsorber
  Arms: NucleoCapture Treatment

SUMMARY:
This is a prospective, multinational, multicentre, randomised, parallel-group, open-label study to assess the safety, tolerability and performance of the NucleoCapture extracorporeal apheresis device in the reduction of circulating cell-free DNA (cfDNA)/Neutrophil Extracellular Traps (NETs) in sepsis patients.

DETAILED DESCRIPTION:
This study investigates the safety, tolerability and performance of the NucleoCapture extracorporeal apheresis device in patients with sepsis and respiratory failure. Sepsis is a common condition in hospital settings and is associated with high rates of morbidity and mortality and despite ongoing development in the treatment and supportive care of sepsis, mortality remains considerable.

cfDNA/NET therapeutic apheresis with NucleoCapture is indicated for the treatment of sepsis and for the treatment/prevention of septic shock. Participants will be randomised to receive either standard of care (SOC) or SOC plus NucleoCapture treatment, SOC will be according to the current guidelines described by the Surviving Sepsis Campaign: international guidelines for the management of sepsis and septic shock. Participants in the SOC plus NucleoCapture arm will receive one treatment session with NucleoCapture per day, for the first three days. Each treatment session with NucleoCapture will last for up 6 hours, aiming to treat 4.5 plasma volumes. Treatment sessions with NucleoCapture treating less than 3.5 plasma volumes will be counted as incomplete and the treatment session will be repeated on the following day, up to day 5 maximum.

Assessments and tests will take place for all participants whilst in Intensive Care Unit (ICU) on days 1 to 5, day 7, day 14, day 21 and day 28. Participants transferred to ward-based care before day 28 will receive no further study assessment visits from the point of transfer to ward-based care, apart from day 28 in which participants will receive a final study assessment visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-75
* Proven or suspected respiratory sepsis aetiology
* Acute respiratory failure currently requiring invasive mechanical ventilation for not more than 48 hours duration
* Horowitz Index for Lung Function (Pa02/Fi02 Ratio) ≤200mmHg or ≤26.6kPa
* Sequential organ failure assessment score (SOFA) ≥4 and ≤ 14
* Have provided written informed consent or consent is given by the patient's legally designated representative or an independent physician (if possible, according to local law).

Exclusion Criteria:

* Expected duration of invasive mechanical ventilation less than 48 hours
* The use of other non-routine extracorporeal sepsis treatments such as very high flux renal replacement therapy (>60ml/kg/h total exchange), use of high cut off filters or other non-routine extracorporeal treatment columns such as Cytosorb, Toramyxcin, etc).
* Presence of severe multiple organ failure at the point of enrolment as evidenced by:

  * Severe refractory vasoplegic failure

    * Norepinephrine dose > 0.60 μg/kg/min
    * Use of epinephrine
  * Concomitant cardiogenic shock, clinically suspected or CI<2.2 if measured

    * Use of dobutamine, epinephrine, phosphodiesterase inhibitors or levosimendan
  * Coagulopathy as defined by platelet count <50
* Calculated Plasma Volume greater than 5000ml as determined by an estimation of total blood volume (according to Nadler's formula, incorporating height, weight and sex) multiplied by (1- Haematocrit). A total blood volume calculator is available at https://www.omnicalculator.com/health/blood-volume
* Long term oxygen therapy or home oxygen use
* Liver cirrhosis (histologically proven or clinically suspected)
* Active bleeding
* Citrate intolerance if citrate is required for therapeutic apheresis
* Heparin allergy if heparin is required for therapeutic apheresis
* Metastatic disease with life expectancy of <12 months and ECOG score of at least 2
* Haematological malignancy if not in remission
* Solid organ transplant and concomitant use of immunosuppression
* Dialysis dependent Chronic Kidney Disease (CKD Stage 5-D)
* Prior use of cardiopulmonary resuscitation (CPR) in index admission
* Requirement for extracorporeal membrane oxygenation (ECMO)
* Patient expected to die within 48 hours of admission to ICU
* Known allergy to components of NucleoCapture
* Current Participation in another interventional clinical trial
* Pregnancy (as established by the presence of beta human chorionic gonadotropin in urine or blood)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-05-05 (Estimated); Study Completion 2027-05-28 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the NucleoCapture column reduces the amount of cfDNA/NETs in the plasma of participants with sepsis and respiratory failure | Within 6 hours from the baseline (pre-column) plasma
  The mean reduction of an expected ≥50% of the net amount of cfDNA/NETs across the NucleoCapture column at the end of each NuceoCapture treatment session

SECONDARY OUTCOMES:
Mean reduction in circulating cfDNA/NETs measured by circulating blood levels of nucleosomes (H.3.1) | Before and after treatment with the NucleoCapture column and at the start and end of a 6 hour period in the SOC treatment arm
  Mean relative reduction of circulating blood cfDNA/NETs at the end of a complete treatment session with NucleoCapture compared to the change in the mean levels of cfDNA/NETs over a 6 hour period in the SOC treatment arm
The clinical benefit of the NucleoCapture column in participants with sepsis and respiratory failure | From date of randomisation to day 21 for organ support and day 28 for survival
  Change in organ support and survival

OTHER OUTCOMES:
The biological efficacy and performance of NucleoCapture will be assessed using routine biomarkers | At baseline, days 1 to 5, day 7 and day 14
  Routine organ function, haematology, coagulation and inflammation biomarkers will be measured
The biological efficacy and performance of NucleoCapture will be assessed using non-routine biomarkers | At baseline, days 1 to 5, day 7 and day 14
  Non-routine biomarkers of inflammation and coagulation will be measured
Device handling and usability | Day 1 up to day 5
  Usability and handling of the device will be assessed in the intervention arm

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Aswani, Principal Investigator — Santersus AG
Locations (9):
- Germany (3):
  - University of Bonn, Bonn
  - Technical University Dresden, Dresden
  - Hannover Medical School, Hannover
- University of Zurich, Zurich, Switzerland
- United Kingdom (5):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Royal Infirmary of Edinburgh, Edinburgh
  - Liverpool University Hospital, Liverpool
  - Guy's and St Thomas' Hospital, London
  - University College London, London

IPD SHARING:
Plan to Share IPD: No